CLINICAL TRIAL: NCT02701387
Title: The Effect of Implant Macro-Thread Design on Implant Stability in the Early Post-Operative Period: A Randomized, Controlled Pilot Study
Brief Title: Effect of Implant Thread Design on Implant Stability Quotient (ISQ) in Early Healing Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Perry R Klokkevold, DDS, MS, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLA Megagen AnyRidge ISQ
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Partial Edentulism
Keywords: bone implant interaction; implant stability; resonance frequency analysis (RFA); implant stability quotient (ISQ)
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AnyRidge Implant (Experimental): Experimental implant (Megagen AnyRidge dental implant) placed in a healed edentulous site to replace a missing tooth.
  Interventions: Device: Megagen AnyRidge dental implant
- EZ Plus Implant (Active Comparator): Comparative implant (Megagen EZ Plus dental implant) placed in a healed edentulous site to replace a missing tooth.
  Interventions: Device: Megagen EZ Plus dental implant

INTERVENTIONS:
Device: Megagen AnyRidge dental implant — AnyRidge is an approved dental implant with a knife edge, thin thread design available in various thread widths (depth).
  Arms: AnyRidge Implant
Device: Megagen EZ Plus dental implant — EZ Plus is an approved dental implant with a standard thread design (width and depth) and that is comparable to many other dental implants currently available on the market.
  Arms: EZ Plus Implant

SUMMARY:
The purpose of this study is to determine whether implant thread design impacts bone remodeling and/or dental implant stability in the early healing period.

The population of this study will consist of a group of subjects who are interested in replacing two or more missing teeth with dental implants. All implant sites will be healed and not require bone augmentation for the placement of a standard 4 mm diameter implant. Subjects first will undergo a brief screening exam. If accepted, comprehensive oral exam will be completed. Subsequently, enrolled subjects will be scheduled for dental surgery to place the implant(s). Subjects will return weekly for the first 8 weeks after placement for a brief post-operative appointment in order to conduct measurements for the study.

DETAILED DESCRIPTION:
Study Design/Sample. This study will be a prospective cohort study. The study sample will be derived from patients presenting to the study site in need of at least two dental implants and who satisfy the criteria listed below. The study site for this project will be University of California, Los Angeles (UCLA) Postgraduate Periodontics and Implant Surgery Clinic. Implant surgeries will be performed by postgraduate periodontal residents of this program. Any resident involved in this study will have had previous experience in placing dental implants. Also, the residents will be, at all times, under the supervision of attending faculty with extensive experience in dental implant surgery.

The implants to be used in this study are Easy (EZ) Plus and AnyRidge. Both implants are manufactured by Megagen Implants United Kingdom (UK) and are currently on the market. The EZ Plus fixture features a "conventional" macroscopic thread design with self-tapping threads with four cutting edges. The AnyRidge fixture features a unique knife-edge thread design. The company claims this thread design results in "maximum bone to implant contact (BIC), maximized compressive force resistance and minimized shear force production," thereby preventing a drop in stability in the immediate post-placement healing period. Both fixtures are manufactured with the same material and surface (Super Resorbable Blast Media (RBM) Surface). Therefore, the only difference between the two implants is the macroscopic thread design.

Potential implant sites will be evaluated clinically and radiographically to determine the amount and location of available bone for the placement of dental implant(s). Implant sites are deemed appropriate when bone height (crest of ridge to vital anatomic structure such as the mandibular nerve canal) is equal to or greater than the length of the proposed implant plus 2+mm (margin of safety). In the case of locations without vital anatomic structures, the bone height may be equal to the length of the implant. The width of available bone should be at least 3mm greater in diameter than the proposed implant (i.e. at least 1.5mm of bone on all sides of the implant). Thus, a 4mm diameter implant requires a minimum of 7mm width of bone (anterior-posterior and mesial-distal). Finally, two implants may be placed next to one another when the available bone meets the above criteria for two implants (i.e. two 4mm implants require 14mm of bone with 3mm bone between the implants). As an example of the required minimum measurement for two 4mm implants: (1.5mm + 4mm + 1.5mm) + (1.5mm + 4mm + 1.5mm) = 14mm.

Following an appropriate medical evaluation and comprehensive clinical and radiographic examination, treatment for patients selected for this study will be executed according to the following standardized protocol:

1. Alginate or polyvinyl siloxane (PVS) impression of maxillary and/or mandibular arch
2. Fabrication of a radiographic stent using [materials]
3. Cone Beam Computed Tomography (CBCT) scan (J. Morita, 3D Accuitomo 170) of implant site
4. Fabrication of a computer generated guide using (Megagen or Anatomage InVivo 5 implant planning software)
5. Guided surgical placement of dental implant(s) using (Megagen or Anatomage Surgical Guide) with a one-stage approach. The implant size (diameter and length) will be determined individually based on usual parameters of implant selection.
6. Resonance frequency analysis measurements using (Osstell ISQ meter). These measurements are done by connecting a metal post to the top of the dental implant. This post is then connected to the ISQ meter which resonates at a certain frequency and provides the operator with a numerical value correlating to the stability of the implant. Taking these measurements does not harm the patient or the implant in any way. This technology is in widespread use among clinicians as a means of assessing implant stability.

   1. Immediately after placement
   2. Weekly for the first eight weeks

Measuring implant stability quotient (ISQ) using resonance frequency analysis (RFA) is not considered "standard of care" but as data from this technology is collected, analyzed and published, it is conceivable that it may become a standard of care procedure for dental implants (e.g. at the time of implant placement and after a period of healing just prior to placing an implant restoration in function).

Whenever it is clinically acceptable to do so, patients needing more than one implant will receive both the EZ Plus implant and the AnyRidge implant, thereby serving as internal controls. Implants may be placed adjacent to one another and/or adjacent to remaining natural teeth. No sites will receive any type of implant-supported provisional restoration. All implants will receive a short healing abutment that protrudes through the gingiva but remains out of occlusion.

For patients requiring two implants, the type of the implant placed in the first site will be determined by a coin flip. The second implant placed will automatically be the other type. For patients requiring three or more implants, an analogous process will occur (i.e. coin flip to decide the first, third, etc. implant type; the second, fourth, etc. will automatically be of the other type).

Data Collection. Data will be collected in a standardized, coded fashion. Data collection sheets will be stored in a locked file cabinet at the study site. Data will be entered into a password-protected database. At the completion of the study including analysis and publication, the data sheets will be destroyed.

Limitations. The limitations of this study include examining only two macroscopic implant designs. Conclusions drawn from this study may guide future research projects with the ultimate goal of minimizing or eliminating the transient drop in implant stability following implant placement and establishing protocols for immediately loaded prostheses based in resonance frequency analysis.

ELIGIBILITY:
Inclusion Criteria:

* Missing two or more teeth with a desire to receive an implant-supported or implant-assisted tooth replacement
* Healed maxillary or mandibular edentulous site for implant placement
* Sufficient bone volume in the site to allow implant placement without the need for bone augmentation

Exclusion Criteria:

* Systemic disease, medication, or habit known to negatively influence bone healing and/or dental implant success

  * Poorly controlled diabetes (HbA1c > 8%)
  * History of bisphosphonate use
  * History of head & neck radiation therapy affecting the proposed implant site
  * History of smoking >10 cigarettes/day (within past 12 months)
  * Current use of medications that adversely affect healing (e.g. corticosteroids, chemotherapeutic drugs)
  * Immune compromised condition (resulting from disease or treatment)
* Insufficient bone volume for dental implant placement
* Otherwise contraindicated to undergo periodontal / oral / implant surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry R Klokkevold, DDS, MS, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Patients presenting to the study site in need of at least two dental implants received one of each implant type: Easy (EZ) Plus and AnyRidge (AR).
Period: Overall Study
Arm/Group | All Participants
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients presenting to the study site in need of at least two dental implants received one of each implant type: Easy (EZ) Plus and AnyRidge (AR).
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 60.4 [47 to 72]
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Implant Stability Quotient (ISQ) Value as a Measure of Implant Stability in Bone
Description: Implant Stability Quotient (ISQ) is a scale from 1 to 100, to quantify implant stability in bone (higher values mean higher stability). ISQ numerical values are generated by applying resonance frequency analysis (RFA) or sound waves through a specialized peg attached to the implant. Data were combined to reduce the number of intervals for analysis purposes. Data from intervals were combined as follows:
  Tr0 = T0 (baseline) Tr1 = Average of follow-up week 1 (T1) and follow-up week 2 (T2) Tr2 = Average of follow-up week 3 (T3) and follow-up week 4 (T4) Tr3 = Average of follow-up week 5 (T5) and follow-up week 6 (T6) Tr4 = Average of follow-up week 7 (T7) and follow-up week 8 (T8)
Time Frame: Baseline (T0) and weekly thereafter for 8 weeks (T1-T8)
Population: Seven participants, each missing at least two posterior teeth in the same arch, were enrolled, resulting in 10 matched pairs for analysis. Outcome was assessed per implant, not per individual participant;
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: implants
Arm/Group | AnyRidge Implant | EZ Plus Implant
Number analyzed (Participants) | 7 | 7
Number analyzed (implants) | 10 | 10
units on a scale
  T0 | 79.6 (1.61) | 80.1 (1.37)
  T1 | 79.7 (1.58) | 79.7 (1.31)
  T2 | 80.0 (1.26) | 79.2 (1.29)
  T3 | 80.1 (0.81) | 78.3 (1.41)
  T4 | 80.3 (0.75) | 77.5 (2.03)
  T5 | 80.3 (0.75) | 77.4 (2.41)
  T6 | 80.2 (0.85) | 77.3 (2.70)
  T7 | 80.4 (0.77) | 77.3 (2.74)
  T8 | 80.6 (0.71) | 77.1 (2.73)
Statistical Analysis 1: Comparison: AnyRidge Implant vs EZ Plus Implant; Comparison of ISQ over time. Due to the high number of intervals (T0-T8) relative to the number of observations, data were combined for analysis purposes into 5 comparable intervals as follows: Baseline (T0, unchanged); Tr1=Average of follow-up weeks T1 and T2, Tr2=Average of follow-up weeks T3 and T4; Tr3=Average of follow-up weeks T5 and T6; Tr4=Average of follow-up weeks T7 and T8; Test type: Superiority or Other; p < 0.01, nonparametric for longitudinal — A 2-factor (implant type x time interval) nonparametric analysis for longitudinal data (Brunner et al. 2002) was used to compare test and control implants across time (baseline + four intervals). The R package "nparLD" was used (Noguchi et al. 2012)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes